CLINICAL TRIAL: NCT01819610
Title: A Single Arm, Open Label Study to Compare the Pharmacokinetics, Safety, and Efficacy of SPRIX (Intranasal Ketorolac Tromethamine) in 12 to 17 Year Old Patients vs. Adult Patients (18-64 Years) Undergoing Open Surgical Procedures
Brief Title: Pharmacokinetics, Safety, and Efficacy of SPRIX in 12 to 17 Year Old Patients vs. Adult Patients Undergoing Open Surgical Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1SPR11001
Record Dates: First submitted 2013-02-25; First posted 2013-03-27 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Pain
Keywords: Postoperative pain management
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPRIX (Experimental): Subjects will be administered open label SPRIX according to subject weight.
  Interventions: Drug: SPRIX

INTERVENTIONS:
Drug: SPRIX
  Other Names: SPRIX (intranasal ketorolac tromethemine)

SUMMARY:
A SPRIX trial in pediatric subjects vs. adults undergoing open surgical procedures resulting in at least a moderate pain level. Subjects will receive SPRIX and blood samples will be collected for pharmacokinetic (PK) assessment. Subjects will also be assessed on the safety and efficacy of SPRIX.

DETAILED DESCRIPTION:
This is a study of intranasal (IN) ketorolac tromethamine (SPRIX) in pediatric subjects age 12-17 years vs. adults ages 18-64 years undergoing open surgical procedures that are expected to result in at least a moderate level of pain (i.e., 40 or above on a 0-100 Visual Analog Scale (VAS) in which 0 is no pain and 100 is the worst pain imaginable). Following surgery subjects will receive their 1st dose of SPRIX, if and when pain reaches a VAS of 40 or more, followed by SPRIX administration every 6 hours. Blood samples for PK assessment will then be collected for PK assessment pre-dose, at 0.25, 0.5, 0.75, 1, 2, and 4 hours after the first dose, at 6 hours (immediately before the 2nd dose), and immediately before each of the next several subsequent q6h doses up to the dose to be administered on the morning of post-operative day 2. Blood samples will then be collected at 1, 2, 4, 6, 8, 12, and 24 hours after receiving the morning dose on day 2 (i.e., last blood sample for PK will be collected on the morning of post-operative day 3). Pain intensity (PI) will be assessed using the 0-100 VAS at 0.5, 1, 2, 4, and 6 hours post dose, at 2 hours after the 2nd dose, and then immediately prior to each dose at 12, 18, and 24 hours from baseline. Patients may elect to continue taking SPRIX for a total of 5 days with daily assessments of pain intensity using a diary. A final follow-up phone interview will be conducted 14 days after the final dose of study drug. Thus, each subject's study participation will consist of a screening visit, a treatment/assessment period of up to 5 days, and a follow-up interview.

ELIGIBILITY:
Inclusion Criteria:

* Male of female patients age 12-64 years.
* Undergoing an open surgical procedure expected to result in at least moderate pain (at least 40 on 0-100 VAS).
* Body mass index (BMI)≤ 95th percentile for age.
* Surgical procedures that would allow the subject to likely remain in the hospital until the morning of post-operative day 3 (to complete PK sample collection).
* Willing and able to complete the study procedures and pain scales and to communicate meaningfully with the study personnel (with parental assistance if pediatric).
* In generally good health and capable of undergoing surgery.
* Females at risk of pregnancy were to use an acceptable form of birth control and have a negative serum or urine pregnancy test.
* Willing to refrain from use of non-study analgesics for the duration of the study, from the day of surgery up to post-operative day 4.
* Assents to participation (if pediatric) and his/her parent or guardian is willing and able to sign the informed consent approved by the IRB. Consents to participation and willing and able to sign the informed consent approved by the IRB if adult.

Exclusion Criteria:

* Surgical procedure performed exclusively by laparoscopy.
* Known allergy or sensitivity to ketorolac, ethylene diamine tetraacetic acid (EDTA), or any nonsteroidal anti-inflammatory drug (NSAID).
* Prior nasal-septal injury or surgery.
* History of peptic ulcer, gastro-esophageal reflux, or gastrointestinal bleeding.
* History of advanced renal impairment or a risk for renal failure due to volume depletion.
* Clinically significant (in the Investigator's opinion) laboratory test value outside the normal range.
* Use of either (a) oxycodone at a dose of 30 mg/day or more or (b) an equivalent dose of another opioid analgesic for a total of more than half of the days during the preceding month.
* The patient requires regular use (daily use in at least 25 days per month) in the 3 months prior to surgery of NSAIDs, COX2 inhibitors, tramadol, or acetaminophen at a daily dose of more than 2 g for the management of pain.
* Contraindication to the use of morphine, general anesthetics, bupivacaine, ropivacaine, lidocaine, other local anesthetics, muscle relaxants, hydrocodone, ondansetron, or acetaminophen (eg, significant history of allergic reactions or intolerance to these or related substances).
* Known bleeding diathesis or other disorder or current use of agents affecting coagulation. Deep venous thrombosis prophylaxis of the surgeon's choice is permitted postoperatively.
* Current use of CNS active drugs such as benzodiazepines, tricyclic antidepressants, or SSRIs for pain. These drugs are permitted for non-pain indications if the dose has been stable for at least 30 days. The use of lorazepam and other sleep medications, except those containing analgesic properties, are permitted.
* Current diabetes mellitus and HbA1C > 9.5 or a history of prolonged uncontrolled diabetes.
* Use of an antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days.
* Any medical condition that in the investigator's opinion could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including active infection.
* History of drug, prescription medicine, or alcohol abuse that would interfere with the subject's safety or the assessments of efficacy in this trial, in the judgement of the investigator.
* History of nasal mucosal damage or active seasonal allergies, nasal congestion, or upper respiratory tract infection sufficient to interfere with intranasal drug delivery.
* Administration of an investigational product within 3 months prior to the first dose of study drug, or scheduled to receive an investigational product, while participating in the study.
* Use of Toradol (ketorolac tromethamine) in any formulation within the past 30 days prior to study entry and throughout study participation.

Ages: 12 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2013-02; Primary Completion 2014-03 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose & .25, .5, .75, 1, 2, 4 hrs after the dose @ 6 hrs & prior to each ensuing dose until morning of post-operative Day 2. After a single dose on the morning of post-operative Day 2 further PK samples will be collected @ 1, 2, 4, 6, 8, 12, & 24 hrs
Ctrough | Pre-dose & .25, .5, .75, 1, 2, 4 hrs after the dose @ 6 hrs & prior to each ensuing dose until morning of post-operative Day 2. After a single dose on the morning of post-operative Day 2 further PK samples will be collected @ 1, 2, 4, 6, 8, 12, & 24 hrs
tmax | Pre-dose & .25, .5, .75, 1, 2, 4 hrs after the dose @ 6 hrs & prior to each ensuing dose until morning of post-operative Day 2. After a single dose on the morning of post-operative Day 2 further PK samples will be collected @ 1, 2, 4, 6, 8, 12, & 24 hrs

CONTACTS AND LOCATIONS:
Overall Officials: David Bregman, M.D, Ph.D., Study Director — American Regent, Inc.
Locations (1):
- Luitpold Pharmaceuticals, Inc., Norristown, Pennsylvania, United States